CLINICAL TRIAL: NCT06297629
Title: A Phase I/II Trial to Assess the Efficacy and Toxicity of ASTX727 (Oral Decitabine/Cedazuridine) for the Treatment of Hematological Neoplasms After Allogeneic Stem Cell Transplantation
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Abandoned
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Astex Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0636; NCI-2024-01689 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2024-02-21; First posted 2024-03-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-04

CONDITIONS: Allogeneic Stem Cell Transplantation
MeSH Terms: interventions — decitabine and cedazuridine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): If participants test positive for minimal residual disease (MRD), participants will be enrolled in Group 1. MRD refers to small numbers of cancer cells that remain in the body during or after treatment. Participants in this group will receive ASTX727 and DLI. If participants are enrolled in Group 1, the participant will take ASTX727 on Days 1-4 of each cycle.
  Interventions: Drug: ASTX727; Drug: Donor Lymphocyte Infusion
- Group 2 (Experimental): If participants do not test positive for MRD, you will be enrolled in Group 2. Participants in this group will only receive ASTX727. If participants are enrolled in Group 2, the participant will take ASTX727 on Days 1-3 of each cycle.
  Interventions: Drug: ASTX727

INTERVENTIONS:
Drug: ASTX727 — Given by PO
  Other Names: Inqovi
Drug: Donor Lymphocyte Infusion — Given by Infusion
  Other Names: DLI
  Arms: Group 1

SUMMARY:
To learn if ASTX727 given alone or in combination with donor lymphocyte infusion (DLI) can help to control certain types of hematological neoplasms (blood-based cancers) after a stem cell transplant.

DETAILED DESCRIPTION:
Primary Objectives

* To determine the safety and toxicity of ASTX727 with or without donor lymphocyte infusion (type, frequency, severity of adverse events [AEs] and relationship of AEs to ASTX727) in the study population (cohort #1 and cohort #2).
* To estimate the complete response (CR) rate of ASTX727 with or without donor lymphocyte infusion (DLI) for the eradication of minimal residual disease (MRD) in participants with acute myeloid leukemia (AML) and myelodysplastic syndrome (MDS), after hematopoietic stem cell transplantation (cohort #1).
* Estimate relapse-free survival (RFS) with the use of ASTX727 as maintenance therapy in participants with high-risk AML and MDS after study entry following hematopoietic stem cell transplantation (cohort #2).

Secondary Objectives

* Participants with creatinine clearance 40-60 cc/min at enrollment will be observed and reported for safety and toxicity separately.
* To determine the overall response and response duration in cohort #1, in participants with MRD detected in the post-transplant setting.
* Duration of remission after study entry following allogeneic stem cell transplant for cohort #2.
* To determine incidence of acute and chronic graft versus host disease (GvHD)
* To evaluate overall survival (OS).

Exploratory Objective

* To investigate possible relationships between protein and gene expression signatures/mutation profile and DNA methylation in predicting relapse-free survival time to the ASTX727.
* To gain insight into clinically relevant genomic factors influencing transplant outcomes, especially into the mechanism of relapse after transplant.
* To characterize the composition of different T-cell subsets, and to determine how those correlate with each other and with transplant outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AML and MDS according to World Health Organization (WHO) classification that underwent first or second allogeneic HSCT with either peripheral blood or bone marrow as the source of the hematopoietic stem cells.
* Age 18 to 75 years old.
* High risk patients defined per cohorts as below:
* Cohort #1: AML and MDS patients in morphological remission with persistence or reappearance of MRD by flow cytometry or molecular after allogeneic stem cell transplantation who are beyond day 100 after allogeneic stem cell transplantation.

  * When MRD is detected by flow cytometry, disease level at or above the sensitivity level of the test will be required.
  * MRD level at or above 0.1%.
  * When MRD is detected by molecular testing, disease level at or above the sensitivity level of the test will be required.
  * The limit of detection is 0.01%
* Cohort #2: High risk AML and MDS patients who are in complete remission morphologically with no evidence of minimal residual disease by flow cytometry or cytogenetic or molecular testing within 100 days after allogeneic stem cell transplantation.
* MDS patients:

  * Moderate-high, high or very high-risk groups by International Prognostic Scoring System-Molecular (IPSS-M) classification if classification is available (58).
  * TP53 with biallelic mutations(49).
  * Therapy-related MDS(50).
  * Presence of mutation ASXL1, SRSF2, DNMT3A, RUNX1, U2AF1, TP53, EZH2, STAG2, CBL, NRAS, BCOR ((49, 51-54))
  * Bone marrow blast count 10% or higher prior to allogeneic stem cell transplantation.
* AML patients

  * Cytogenetics and molecular features consistent with adverse risk group by 2017 European LeukemiaNet classification for AML(55)
  * Presence of MRD by multi-color flow cytometry or cytogenetics or molecular studies by the last bone marrow evaluation prior to HSCT.
  * Primary induction failure defined as absence of complete remission after two different lines of anti-leukemia therapy following diagnosis.
  * Presence of active disease defined as bone marrow blast count >5% but <= 20% at the time of HSCT.
  * Patients transplanted beyond first CR.
  * Therapy-related AML.
  * Overexpression of EVI1 (52)
* All patients in cohort #2:

  * Post-transplant bone marrow consistent with complete remission with no evidence of minimal residual disease by flow-cytometry or cytogenetics or molecular testing.
  * Adequate engraftment within 7 days prior to starting study drug: Absolute neutrophil count (ANC) >/= 1.0 x 109/L without daily use of myeloid growth factor (G-CSF) for at least 7 days; and,platelet >/= 30 x 109/L without platelet transfusion within 1 week.
* ECOG performance status of 0, 1, or 2.
* Creatinine clearance greater or equal than 40 cc/min as defined by the Cockcroft-Gault Equation*.

Males (mL/min) :(140-age) *IBW (kg) / 72*(serum creatinine(mg/dl)) Females (mL/min):0.85*(140-age) *IBW (kg) / 72*(serum creatinine(mg/dl)).

* Serum bilirubin </= 1.5 x upper limit of normal (ULN). Aspartate transaminase (AST) or alanine transaminase (ALT) </= 2.5 x ULN. Alkaline phosphatase </= 2.5 x UL.
* No active bleeding.
* No clinical evidence of life-threatening infection. Capable of understanding the investigational nature, potential risks and benefits of the study, and able to provide valid informed consent.
* Negative serum or urine pregnancy test for women with reproductive potential. The only subjects who will be exempt from this criterion are postmenopausal women (defined as women who have been amenorrheic for > 12 months) or subjects who have been surgically sterilized or otherwise proven sterile.

Females of childbearing potential must refrain from becoming pregnant and commit to either apply highly effective method of birth control (two reliable methods of birth control) or continue abstinence from heterosexual intercourse during study period and for at least 6 months after last dose of ASTX727. Male subjects who are sexually active with a women of childbearing potential (WOCBP) and who have not had vasectomies must be willing to use a barrier method of contraception and refrain from sperm donation from initial study drug until 3 months after last dose of study drug.

Exclusion Criteria:

* Use of any anti-leukemic agents after MRD is documented (note that the use of these anti-leukemic agents given as post-transplant maintenance therapy is allowed in this study, e.g., subcutaneous or oral 5-Azacytidine or FLT3 inhibitors for maintenance, for cohort #1 patients. However, all those agents will be discontinued once the patient enrolls into the current trial for cohort #1.
* Use of any of the following after transplantation and prior to starting study therapy for cohort #2. Anti-leukemic agents given as post-transplant maintenance therapy (e.g., subcutaneous or oral 5-Azacytidine or FLT3 inhibitors for maintenance).
* Overall grade II-IV acute GVHD. However, upon complete resolution of acute GVHD-related symptoms, patients are eligible for enrollment if they are on prednisone 0.5 mg/kg daily dose or lower, tacrolimus, sirolimus and ruxolitinib.
* Chronic GvHD, moderate or severe by NIH criteria.
* Active uncontrolled systemic fungal, bacterial or viral infection. However, patients receiving anti-microbial agents including antibiotics, antiviral and antifungal therapies are allowed if hemodynamically stable.
* Symptomatic or uncontrolled arrhythmias.
* Significant active cardiac disease within the previous 6 months, including:
* New York Hear Association (NYHA) class III or IV congestive heart failure;
* Unstable angina or angina requiring surgical or medical intervention, and/or; Myocardial infarction.
* Known active viral infection with Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV) or Hepatitis C Virus (HCV).

  * Patients with known active hepatitis B virus (HBV) infection will be excluded because of potential effects on immune function and/or drug interactions. However, if a patient has HBV history with an undetectable HBV load by polymerase chain reaction (PCR), no liver-related.

complications, and is on definitive HBV therapy that is not contraindicated on this study, then he/she would be eligible for study.

* Patients with known active hepatitis C virus (HCV) infection will be excluded because of potential effects on immune function and/or drug interactions. However, if a patient with a history of HCV infection has received definitive therapy (and is now HCV viral load negative), or if a patient has a reactive HCV antibody test but has an undetectable viral load by PCR, then he/she would be eligible.
* Patients with known active HIV infection will be excluded out of concern for the drug-drug interaction with venetoclax and highly active antiretroviral therapy (HAART).

  - Prior history of solid tumors other than AML and MDS, unless the subject has been free of the disease for >/= 1 year. However, subjects with the following history/concurrent conditions are allowed:
* Basal or squamous cell carcinoma of the skin;
* Carcinoma in situ of the cervix;
* Carcinoma in situ of the breast;
* Incidental histologic finding of prostate cancer (T1a or T1b using the tumor, node, metastasis [TNM] clinical staging system).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-07-11 (Actual); Study Completion 2024-07-11 (Actual)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Betul Oran, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org